CLINICAL TRIAL: NCT00642681
Title: Evaluation of the Effect of Symptomatic Upper Respiratory Infections on Pharmacological Characteristics of Technosphere®/Insulin in Subjects With Diabetes Mellitus After a Meal Challenge
Brief Title: Effects of URI on Diabetic Subjects Utilizing Technosphere Insulin After a Meal Challenge
Status: Completed | Type: Observational
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MKC-TI-112
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus; Upper Respiratory Infection
MeSH Terms: conditions — Diabetes Mellitus; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: TI Inhalation Powder: Technosphere® Insulin (TI) Inhalation Powder
  Interventions: Drug: Technosphere Insulin

INTERVENTIONS:
Drug: Technosphere Insulin — Technosphere® Insulin (TI) Inhalation Powder, prandial

SUMMARY:
Effect of upper respiratory infection (URI) on diabetic subjects with a meal challenge

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have met the same inclusion criteria as MKC-TI-030
* Clinical diagnosis of URI with in 24 hrs prior to clinic visit and/or day of clinic visit
* At least 3 URI symptoms

Exclusion Criteria:

* Prior participation in MKC-TI-112
* MedHist, PE or lab findings of acute bacterial infection including but not limited to sputum prod., nasal/eye discharge, chest exam abnormalities, CXR findings of pneumonia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who developed symptoms of URI at any point during the MKC-TI-030 trial and were randomized to study treatment of TI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To measure Serum FDKP AUC | 4 Hours

CONTACTS AND LOCATIONS:
Locations (24):
- United States (15):
  - Arizona Research Associates, Tuscon, Arizona
  - Valley Research (Norwood), Fresno, California
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - Private Practice, Decatur, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Cedar-Crosse Research Center, Chicago, Illinois
  - MODEL Clinical Research, Baltimore, Maryland
  - Healthcare Research, Florissant, Missouri
  - Billings Clinic Research Division, Billings, Montana
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - M.E.R.I., New York, New York
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Your Diabetes Endocrine Nutrition Group, Mentor, Ohio
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - Magna Center for Family Medicine, Magna, Utah
- Parkwood Hospital, London, Ontario, Canada
- Russia (8):
  - Kemerovo State Medical Academy of Ministry of Health, Kemerovo, RUS
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - Russian State Medical University City Hospital # 4, Moscow, RUS
  - RAAMS Endocrinology and Diabetology Department, Moscow, RUS
  - Clinical Pharm Dept of Yaroslavl Clin Hospital, Yaroslavl, RUS
  - NHI Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - FSI Principal Military Clinical Hospital n.a. academician N.N. Burdenko of the Ministry of Defense, Moscow